CLINICAL TRIAL: NCT02313623
Title: MR-US Image Fusion Targeted Biopsy for Single-cell Prostate Cancer Research
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1304011902
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Research samples will be placed in separate, de-identified specimen jars. Following each case, investigators on this protocol will provide the de-identified specimen jars to collaborators to perform single-cell analysis. All clinical specimens will be handled by pathology according to existing protocols.
  Processing of the samples will include disassociated into a single cell suspension and culturing the sample. This suspension can be then placed onto a microfluidic device for processing. It is hypothesized that collection of samples in this manner will allow the comparison of molecular profiles with clinically accepted standards to impact prospective research on prostate cancer.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient Scheduled for Prostate Fusion Biopsies: For subjects with scheduled fusion biopsies, we propose a research plan to acquire additional biopsy cores for research purposes without impacting clinical protocol. After acquiring clinically-necessary biopsies, we propose taking an additional research biopsy to establish a matched-pair of clinical and research samples.
  Interventions: Procedure: Prostate Fusion Biopsy

INTERVENTIONS:
Procedure: Prostate Fusion Biopsy — For subjects with scheduled fusion biopsies, we propose a research plan to acquire additional biopsy cores for research purposes without impacting clinical protocol. After acquiring clinically-necessary biopsies, we propose taking an additional research biopsy to establish a matched-pair of clinical and research samples.

SUMMARY:
The investigators hypothesize that this single-cell analysis can be used to evaluate prostate needle-core biopsies prospectively even in non-homogenous samples by providing profiles of proteomic and phenotypic signatures. These profiles will in turn enable better predictions of the malignant progression of prostate cancers in the settings of current clinical practice.

DETAILED DESCRIPTION:
Current approaches for early detection and diagnosis include prostate-specific antigen (PSA) which is a useful, though not specific, biomarker for detecting prostate cancer. The suspected patients will be further sent for digital rectal examination(DRE), in which a doctor inserts a lubricated, gloved finger into the patient's rectum to feel for lumps, enlargements, or areas of hardness that might indicate prostate cancer. However, the only test that can fully confirm the diagnosis of prostate cancer is a biopsy - the removal of small pieces of the prostate for microscopic examination. If cancer is suspected using PSA test and DRE, more than 90% suspected patients choose undergo prostate biopsy. Prostate needle biopsies are routinely done on an outpatient basis and rarely require hospitalization. Markedly, the fine needle biopsy is minimally invasive and has currently been suggested for longitudinal monitoring of highly suspected patients or follow-up therapeutic responses. The large availability of biopsy samples for prostate cancer provides a cornerstone for the proposed patient specimen-based research. The investigators anticipate that comprehensive analysis rather than simple pathological examination of these samples will generate new insights to prostate tumor progression in human.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects that have scheduled Artemis prostate biopsy with defined regions of interest will be included in this study

Exclusion Criteria:

* Any subjects that are unable to provide informed consent will be excluded

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with scheduled Artemis fusion biopsy will be recruited into this study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-07; Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Success Rate of Primary Prostate Cell Culture | 2 years
  how often are primary prostate cancer cells able to be grown in culture

CONTACTS AND LOCATIONS:
Overall Officials: Preston C Sprenkle, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No